CLINICAL TRIAL: NCT00516425
Title: Adjuvant Cytotoxic Chemotherapy In Older Women
Brief Title: Doxorubicin or Epirubicin and Cyclophosphamide in Treating Older Women With Invasive Breast Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charing Cross Hospital (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: UKM-CCH-ACTION; CDR0000561076 (Registry Identifier: PDQ (Physician Data Query)); ICR-CTSU/2006/10004-ACTION; EU-20751; EUDRACT-2005-005721; ISRCTN41708421; BIG-205
Record Dates: First submitted 2007-08-14; First posted 2007-08-15 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2007-09

CONDITIONS: Breast Cancer
Keywords: stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pegfilgrastim; Cyclophosphamide; Doxorubicin; Epirubicin; Spectrometry, Mass, Matrix-Assisted Laser Desorption-Ionization; Chemotherapy, Adjuvant

INTERVENTIONS:
Biological: pegfilgrastim
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: epirubicin hydrochloride
Genetic: proteomic profiling
Other: diagnostic laboratory biomarker analysis
Other: matrix-assisted laser desorption/ionization time of flight mass spectrometry
Other: pharmacological study
Other: surface-enhanced laser desorption/ionization-time of flight mass spectrometry
Procedure: adjuvant therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as doxorubicin, epirubicin, and cyclophosphamide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving combination chemotherapy after surgery may kill any tumor cells that remain after surgery. Sometimes, after surgery, the tumor may not need more treatment until it progresses. In this case, observation may be sufficient. It is not yet known whether giving doxorubicin or epirubicin together with cyclophosphamide is more effective than observation in treating older women with invasive breast cancer.

PURPOSE: This randomized phase III trial is studying doxorubicin or epirubicin and cyclophosphamide to see how well they work compared with observation in treating older women with invasive breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To provide evidence for extending the current standard care in older women with invasive breast carcinoma treated with adjuvant chemotherapy comprising doxorubicin hydrochloride or epirubicin hydrochloride and cyclophosphamide.
* Compare the relapse-free survival interval of these patients treated with adjuvant chemotherapy vs no adjuvant chemotherapy.
* Compare the toxicity of accelerated adjuvant chemotherapy with pegfilgrastim support vs non-accelerated adjuvant chemotherapy.

OUTLINE: This is a multicenter study. Patients are stratified according to participating center and indication for endocrine therapy (yes vs no). Patients are randomized to 1 of 2 arms.

* Arm I (observation): Patients do not receive adjuvant chemotherapy.
* Arm II (adjuvant chemotherapy): Patients are randomized to 1 of 2 chemotherapy regimens.

  * Accelerated adjuvant chemotherapy: Patients receive doxorubicin hydrochloride and cyclophosphamide (AC) OR epirubicin hydrochloride and cyclophosphamide (EC) on day 1 and pegfilgrastim on day 2. Treatment repeats every 2 weeks for 4 courses in the absence of disease progression or unacceptable toxicity.
  * Non-accelerated adjuvant chemotherapy: Patients receive AC or EC on day 1. Treatment repeats every 3 weeks for 4 courses in the absence of disease progression or unacceptable toxicity.

Patients undergo tumor tissue and blood sample collection for biological, pharmacological, and proteomic studies. Samples are initially used to establish a resource of materials available for different research groups. Samples are also analyzed using SELDI or MALDI-ToF technology to identify biological profiles that correlate with prognosis or predict response to treatment.

Quality of life is assessed at baseline, 6 weeks, 1 month, 6 months, 9 months, 12 months, 18 months, and 24 months.

After completion of study treatment, patients are followed every 6 months for 2 years and then annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed invasive breast carcinoma
* Primary operable breast cancer that was surgically treated by wide local excision or mastectomy with clear margins (> 1 mm apart from deep margin if full thickness resection)

  * No more than 8 weeks since prior definitive surgery
* Early-stage disease with no evidence of metastases clinically or on routine staging investigations

  * No T4 and/or N3 disease
* Prior axillary staging required, including 1 of the following:

  * Sentinel node biopsy
  * Axillary sampling or clearance

    * All node-positive patients must have had axillary clearance or radiotherapy to the axilla
* Must be at high risk of relapse within 5 years (risk factors evaluated at clinician's discretion)
* No other invasive breast cancer, systemically treated ductal carcinoma in situ (DCIS), or solid tumor within the past 5 years
* No prior hematologic malignancy or melanoma
* Hormone receptor status:

  * Estrogen receptor (ER)- or progesterone receptor (PR)-negative OR ER/PR-weakly positive (e.g., Allred/Quick score ≤ 5 OR H score ≤ 100)

PATIENT CHARACTERISTICS:

* Female
* Postmenopausal
* Performance status 0-1
* Hemoglobin > 9 g/dL
* WBC > 3,000/mm³
* Platelet count > 100,000/mm³
* Bilirubin normal (unless known Gilbert's disease is present)
* Albumin normal
* AST and ALT ≤ 1.5 x upper limit of normal (ULN)
* Creatinine ≤ 1.5 x ULN
* Creatinine clearance > 50 mL/min
* No active or uncontrolled infection
* Must be available for routine long-term hospital follow-up
* Must have normal cardiac function and no significant cardiac disease by ECHO or MUGA

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 4 weeks since prior preoperative endocrine therapy
* No prior systemic therapy for this breast cancer or mantle radiotherapy
* No prior breast-conserving surgery in which there is a contraindication for, or decline of postoperative radiotherapy
* No concurrent hormone replacement therapy (HRT)

Min Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2007-01

PRIMARY OUTCOMES:
Relapse-free interval
Physical, functional, and breast cancer concerns as measured by the Trial Outcome Index (TOI)
Total FACT-AN score
Total FACT-F score

SECONDARY OUTCOMES:
Disease-free survival
Overall survival
Cause-specific survival
Distant disease-free survival
Safety and tolerability (overall and for each treatment schedule)
Treatment compliance (overall and for each treatment schedule)
Quality of life
Total FACT-B score
Individual subscales on activities of daily living

CONTACTS AND LOCATIONS:
Overall Officials: Robert C.F. Leonard, MD, BS, MB, Principal Investigator — Charing Cross Hospital
Locations (2):
- United Kingdom (2):
  - Charing Cross Hospital, London, England
  - Southend University Hospital NHS Foundation Trust, Westcliff-on-Sea, England